CLINICAL TRIAL: NCT05598840
Title: Randomized Clinical Trial to Assess the Efficacy of a Mobile Application to Help in Weight Loss Before Bariatric Surgery: the VAMOS Project (Virtual Accompaniment for Morbid Obesity Surgery)
Brief Title: Efficacy of a Mobile Application to Help in Weight Loss Before Bariatric Surgery
Acronym: VAMOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Javier Osorio, Chief of Bariatric and Metabolic surgical Unit, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUB-VAMOS
Record Dates: First submitted 2022-09-23; First posted 2022-10-28 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Morbid Obesity; Weight Loss
Keywords: Mobile APP; Obesity; R-en-Y gastric bypass; Preoperative weight loss
MeSH Terms: conditions — Obesity, Morbid; Weight Loss; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APP group (Experimental): Four months before surgery, the C4T APP, in addition to standard protocol, will be provided to all the patients randomized in the APP group.
  Interventions: Other: Care for today Mobile Application
- Normal VLCD (Very Low Calory Diet) group (Active Comparator): Normal preoperative standard protocol will be provided to all the patients randomized in the normal group.
  Interventions: Other: Care for today Mobile Application

INTERVENTIONS:
Other: Care for today Mobile Application — C4T (Care for Today) Education is a digital application (app) designed to offer quality educational materials.
  The APP will be provided to the patients in the outpatient centre four months before surgery. Patients will be able to download the APP using a QR code that will be provided during the visit. They'll realize the download immediately or at home, in both cases a detailed explication of how to use the APP and its contents will be provided using an example version.

SUMMARY:
The present randomized clinical trial aims to prove the safety and efficacy of an interactive mobile application (Care4Today®) to obtain sufficient weight loss and empower patients with morbid obesity before being submitted to a gastric by-pass.

DETAILED DESCRIPTION:
Morbid obesity is considered the great epidemic of our century. It is regarded as the first non-traumatic cause of death in the western population and it is also progressively beginning to affect developing countries. The latest epidemiological studies estimate that in Spain more than 15% of the population has overweight and about 5% has morbid obesity.

Obesity treatment is multidisciplinary, from lifestyle and dietary changes to surgery. Amongst the different available treatments, bariatric surgery is the only cost-effective in patients with morbid obesity. Bariatric surgery provides better results compared to both pharmacological treatments (which are less available and less effective) and lifestyle changes. Furthermore, as well as weight loss, it guarantees a better control of comorbidities, reducing the risk of cardiovascular disease, morbidity and mortality, improving quality of life.

Although surgery is the best treatment option, patient commitment is necessary to achieve satisfactory results. Obtaining patient's comprehension of the importance of healthy lifestyle and equilibrated diet alongside with surgical information is generally difficult. Patient's concern needs to be constantly stressed out. The ongoing protocols that include preoperative meetings with surgeons, endocrinologists and nutritionists have been proved as insufficient, especially during the Covid-19 pandemic, when presential visits were reduced or cancelled.

Preoperative optimization with a healthy lifestyle and a balanced diet few months before surgery potentially reduce intraoperative complications alongside with postoperative morbidity and mortality. Level of physical activity, diet and psychological stability could affect surgery's outcome for example reducing liver volume (up to 20%) and mesenteric fat. Also, an improvement in patient's preoperative satisfaction, anxiety and commitment to surgery have been suggested. Their impact on postoperative outcomes is unclear. There is lack of consensus on a standardized preoperative approach and goals. Many health care professionals worldwide strongly believe that preoperative optimization has an important impact on postoperative outcomes, but the evidence supporting this belief is mixed and most often retrospective. Although a positive relationship between self-monitoring behaviors (such as daily food intake diaries and regular self-weighing) and weight loss has been proved, additional instruction and behavioral intervention are needed. Besides weight loss, other factors such as adherence to self-monitoring of weight, recording food intake, increased physical activity could influence postoperative outcomes.

Even though official guidelines for an enhanced recovery (ERAS, Enhanced Recovery After Surgery) in bariatric surgery recommend patient information, education, counseling and preoperative weight loss, the efficacy of these measures has not been proved.

Technological development is an important resource that could help improving communications between patients and health care professionals. Nowadays, the use of a smartphone is widely integrated in daily life of most people. The number of smartphones used is constantly increasing every year. In 2016, there were more than seven billion users worldwide. The worldwide fast widespread of mobile technology in the last 15 years led to an expansion of the applications (APP) market. To date, the biggest APP market are 'Google Play' (Android), 'App store' (Apple) and 'Blackberry World' (Blackberry).

This technological revolution has progressively affected the health world. An increasing number of medical APP have been designed in the last years, few directly managed from health care providers from public or private centers. The Mobile Health APP could led to a simpler, real-time connection between patients and health care professionals alongside with a bidirectional data flow and a steadily monitorization of patients' evolution that could obtain a better preoperative follow-up without increasing the costs.

The present randomized clinical trial aims to prove the safety and efficacy of an interactive mobile application (Care4Today®) to obtain sufficient weight loss and empower patients with morbid obesity before being submitted to a gastric by-pass.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 and younger than 65 years who meet criteria to undergo bariatric surgery

BMI between 35 and 50 kg/m2 and indication of one-time surgery

Signing the informed consent of the study

Patient suitable for laparoscopic surgery

Patient who demonstrates accessibility to a smartphone and basic digital competence

Exclusion Criteria:

* Previous bariatric surgery

Two-step surgery

Patient without resources to access the use of a Smartphone or without basic digital competence

Contraindication for surgery

Other surgical procedures associated with the same intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Preoperative weight loss | App will be provided four months before surgery and then preoperative weight loss achieved will be evaluated the day of surgery
  To compare patients' preoperative weight loss after using the C4T APP versus the standard preoperative protocol.

SECONDARY OUTCOMES:
patient information using the APP | App will be provided four months before surgery and patients' information/satisfaction using the APP will be evaluated the day of surgery
  A validated questionnaire will be used to compare patients' information using the APP vs. standard protocol. (10 questions, 1 point each: >6 good information achieved).
patient satisfaction using the APP | App will be provided four months before surgery and patients' information/satisfaction using the APP will be evaluated the day of surgery
  A validated questionnaire (will be used to compare patients' satisfaction using the APP vs. standard protocol. (10 items to evaluate as very poor, poor, correct, good, excellent).
Correlation between preoperative weight loss and early complications | Early complication rate in each group will be evaluated and compared 30 and 90 days postoperative
  Compare complications in the immediate postoperative period (30- and 90-days post-intervention) after the preoperative use of APP vs. standard protocol. Complications will be recorded in our prospective database.
Correlation between preoperative weight loss and Early postoperative weight loss | Patients' weight loss in each group will be evaluated and compared 3 months after surgery
  Compare patients' weight loss 3 months after surgery using the APP vs. standard protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-07-09): https://cdn.clinicaltrials.gov/large-docs/40/NCT05598840/Prot_SAP_ICF_000.pdf